CLINICAL TRIAL: NCT01342354
Title: A Study of Stereotactic Body Radiation Therapy in Patients With Unresected Carcinoma of the Pancreas or Ampulla
Brief Title: Study of Stereotactic Body Radiation Therapy in Patients With Intact Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16866B
Record Dates: First submitted 2011-04-15; First posted 2011-04-27 (Estimated); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Stereotactic Radiation
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Stereotactic Radiation: 10 Gy x3 (Experimental): Level 1 - SBRT 10Gy in three doses over ten days (total 30 Gy).
  Interventions: Radiation: Stereotactic Radiation 10 Gy
- Stereotactic Radiation: 12.5 Gy x3 (Experimental): Level 2 - SBRT 12.5Gy in three doses over ten days (total 37.5 Gy).
  Interventions: Radiation: Stereotactic Radiation 12.5 Gy
- Stereotactic Radiation: 15 Gy x3 (Experimental): Level 3 - SBRT 15Gy in three doses over ten days (total 45 Gy).
  Interventions: Radiation: Stereotactic Radiation 15 Gy

INTERVENTIONS:
Radiation: Stereotactic Radiation 10 Gy — 10 Gy three times over 10 days
  Arms: Stereotactic Radiation: 10 Gy x3
Radiation: Stereotactic Radiation 12.5 Gy — 12.5 Gy three times over 10 days
  Arms: Stereotactic Radiation: 12.5 Gy x3
Radiation: Stereotactic Radiation 15 Gy — 15 Gy three times over 10 days
  Arms: Stereotactic Radiation: 15 Gy x3

SUMMARY:
This purpose of this study is to determine the highest tolerated dose of Stereotactic Body Radiation Therapy (SBRT) and also to determine the appropriate dose for intact pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, unresected cancer of the pancreas or ampulla. The cancer may include any invasive histology (e.g. adenocarcinoma, neuroendocrine carcinoma).
* Patients must have measurable radiographic disease.Patients with previous complete resection are only eligible if there is measurable radiographic disease which is clearly felt to represent locally recurrent disease.
* Patients may receive any number of cycles of chemotherapy prior to treatment with SBRT, but not within 2 weeks of the first fraction of RT.
* Age > or = 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status < or = 2 (Karnofsky > or = 60%)
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Concurrent investigational therapy delivered over the period of treatment or observation (28 days post-RT) for dose limiting toxicity.
* Prior radiation therapy to the abdominal area which would overlap with the proposed area of treatment.
* Pregnancy.
* Primary disease > 7.5 cm in largest diameter as measured by CT or MRI.
* Gross extension of tumor into the lumen of the duodenum.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Use of bevacizumab or vascular endothelial growth factor inhibitor chemotherapy within 3 months before RT or 6 months after RT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-04-14 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2022-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Liauw, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded Patients (n = 2) due to screening failures
Period: Overall Study
Arm/Group | Stereotactic Radiation: 10 Gy x3 | Stereotactic Radiation: 12.5 Gy x3 | Stereotactic Radiation: 15 Gy x3
Started | 3 | 3 | 9
Completed | 3 | 3 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stereotactic Radiation: 10 Gy x3 | Stereotactic Radiation: 12.5 Gy x3 | Stereotactic Radiation: 15 Gy x3 | Total
Number analyzed (Participants) | 3 | 3 | 9 | 15
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 81] | 55 [40 to 62] | 61 [34 to 69] | 61 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 9
  Male | 1 | 1 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 1 | 7 | 10
  Black or African American | 0 | 1 | 2 | 3
  Hispanic or Latino | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (Phase 1)
Description: Side effects will be assessed after 28 days of treatment to determine tolerability of the dose of radiation.
Time Frame: 28 days
Measure: Number; unit: Gy
Groups:
- Stereotactic Radiation: All participants received one course of SBRT
Arm/Group | Stereotactic Radiation
Number analyzed (Participants) | 15
Gy | 45

2. Secondary Outcome: The Number of Patients With Late (>28 Days) Grade 3+ GI Toxicity
Description: Grade 3+ GI late toxicity
Time Frame: 12 months after treatment
Measure: Number; unit: participants
Arm/Group | Stereotactic Radiation: 10 Gy x3 | Stereotactic Radiation: 12.5 Gy x3 | Stereotactic Radiation: 15 Gy x3
Number analyzed (Participants) | 3 | 3 | 9
participants | 2 | 0 | 2

3. Secondary Outcome: Number of Participants With an Improvement in Patient Reported Pain Score Using Visual Analog Scale
Description: Using the visual analog scale, patients rate pain from 1-10 with higher scores indicate greater pain intensity. Improvement in pain is defined as a yes/no response.
Time Frame: 12 months after treatment
Population: Only eight patients of enrolled patients across all dose levels had pain at presentation and were eligible for this secondary outcome of pain response
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiation: 10 Gy x3 | Stereotactic Radiation: 12.5 Gy x3 | Stereotactic Radiation: 15 Gy x3
Number analyzed (Participants) | 3 | 0 | 5
Participants | 3 | 0 | 2

4. Secondary Outcome: Number of Patients Eligible for Surgery to Remove Tumor After Treatment
Time Frame: 12 months after treatment
Measure: Number; unit: participants
Groups:
- Stereotactic Radiation: 15 Gy x3: Level 1 - SBRT 15Gy in three doses over ten days (total 45 Gy).
Arm/Group | Stereotactic Radiation: 10 Gy x3 | Stereotactic Radiation: 12.5 Gy x3 | Stereotactic Radiation: 15 Gy x3
Number analyzed (Participants) | 3 | 3 | 9
participants | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With Local Disease Control
Description: Number of patients with no disease progression as measured by tumor imaging, based on RECIST criteria
Time Frame: 12 months after treatment
Measure: Number; unit: participants
Arm/Group | Stereotactic Radiation: 10 Gy x3 | Stereotactic Radiation: 12.5 Gy x3 | Stereotactic Radiation: 15 Gy x3
Number analyzed (Participants) | 3 | 3 | 9
participants | 3 | 3 | 5

6. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Using FACT-Hepatobiliary (FACT-Hep) Quality of Life Questionnaire.
Description: The Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) is an instrument that assesses health-related quality of life in patients with hepatobiliary cancers. The FACT-Hep consists of the FACT-G, which assesses generic health-related quality of life and concerns, and a validated Hepatobiliary Subscale (HS), which assesses disease-specific issues. Responses are on a 5 point Likert-type scale; items are summed to generate scores, with higher scores indicating better QOL (possible range of total score = 0-180).
Time Frame: 12 months after treatment
Population: This measure was added to the study protocol when accrual for the third cohort began and thus was only assessed in the third (15 Gy x3) cohort. Among this cohort, baseline data was only collected for 5 patients and only 1 of these patients had 12 month data, which was optional, and that is what is summarized here.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stereotactic Radiation: 10 Gy x3 | Stereotactic Radiation: 12.5 Gy x3 | Stereotactic Radiation: 15 Gy x3
Number analyzed (Participants) | 0 | 0 | 5
score on a scale
  Baseline |  |  | 142 (24)
  12 months: number analyzed (Participants) | 0 | 0 | 1
  12 months |  |  | 157 (0)

ADVERSE EVENTS:
Time Frame: Adverse events as specified in the protocol to meet the definition of dose-limiting toxicity or acute adverse events were monitored for only one month. Serious adverse events ( late GI toxicity) were followed for up to 12 months after treatment. All-cause mortality was assessed over a longer period, which in this case was until death for all enrolled patients and up to 8 years.
Arm/Group | Stereotactic Radiation: 10 Gy x3 | Stereotactic Radiation: 12.5 Gy x3 | Stereotactic Radiation: 15 Gy x3
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 9/9
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 2/9
Other Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Radiation: 10 Gy x3 (N=3) | Stereotactic Radiation: 12.5 Gy x3 (N=3) | Stereotactic Radiation: 15 Gy x3 (N=9)
Gastrointestinal bleeding (Gastrointestinal disorders) | 2 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic Radiation: 10 Gy x3 (N=3) | Stereotactic Radiation: 12.5 Gy x3 (N=3) | Stereotactic Radiation: 15 Gy x3 (N=9)
Nausea (Gastrointestinal disorders) | 1 | 3 | 4
Fatigue (General disorders) | 0 | 1 | 5
Gastrointestinal bleeding (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT01342354/Prot_SAP_000.pdf